CLINICAL TRIAL: NCT00683371
Title: Microarray Analysis of Sinus Samples From Patients With and Without Chronic Rhinosinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H43796-31316-03
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Maxillary Sinusitis
Keywords: Chronic Rhinosinusitis; Sinus Disease; Allergy; Maxillary Sinus; Microarray
MeSH Terms: conditions — Maxillary Sinusitis; Paranasal Sinus Diseases; Hypersensitivity | interventions — Specimen Handling

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 10 patients with chronic rhinosinusitis will have three specimens collected from the maxillary sinus during surgery
  Interventions: Procedure: Specimen collection
- 2 (Placebo Comparator): 10 patients without sinus disease will have three specimens collected from the maxillary sinus during surgery.
  Interventions: Procedure: Specimen collection

INTERVENTIONS:
Procedure: Specimen collection — 10 patients with chronic rhinosinusitis will have three specimens collected from the maxillary sinus during surgery. The sinus mucosa, sinus mucus and a saline lavage will be collected. The three samples will then be analyzed with microarrays looking for bacteria, fungi, and viruses.
  Arms: 1
Procedure: Specimen collection — 10 patients without sinus disease will have three specimens collected from the maxillary sinus during surgery. The sinus mucosa, sinus mucus and a saline lavage will be collected. The three samples will then be analyzed with microarrays looking for bacteria, fungi, and viruses.
  Arms: 2

SUMMARY:
Mucosal biopsies, endoscopically-guided brush samples of mucus, and a saline lavage taken from the maxillary sinuses of ten CRS patients undergoing sinus surgery are analyzed using three microarrays in order to detect bacteria, fungi and viruses. Ten control patients with normal sinuses will have the same samples taken. The hypothesis is that bacterial, fungal, and viral communities present in the maxillary sinus of patients with CRS are significantly different from those patients with healthy sinuses, and that microorganisms identified in patients with or without CRS will differ from previously published data obtained using other techniques.

DETAILED DESCRIPTION:
Mucosal biopsies, endoscopically-guided brush samples of mucus, and a saline lavage taken from the maxillary sinuses of ten CRS patients undergoing sinus surgery are analyzed using three microarrays: 16S rRNA PhyloChip (to detect bacteria), MycoChip (to detect fungi) and ViroChip (to detect viruses). Ten control patients with normal sinuses, as assessed by CT scan and a sinusitis-specific survey, will have the same samples taken. The hypothesis is that bacterial, fungal, and viral communities present in the maxillary sinus of patients with CRS are significantly different from those patients with healthy sinuses, and that microorganisms identified in patients with or without CRS will differ from previously published data obtained using other techniques. Comparing diseased and control flora will provide insight into the relative contribution of each pathogen to CRS and may guide the development of future therapies.

ELIGIBILITY:
Inclusion Criteria (CRS patients):

* History of CRS as defined as symptoms (nasal discharge, nasal obstruction, facial pain and/or hyposmia) for >12 weeks despite therapy.
* Impaired CRS-specific quality of life (SNOT-20 score >1.5).
* Evidence of sinus disease on a CT scan (Lund MacKay score greater than or equal to 10).
* Patients with positive skin or RAST testing to an inhalant allergen and/or aspirin hypersensitivity will be included. Evidence of atopy is not required but will be recorded, along with serum IgE levels, when available.

Inclusion Criteria (Control patients):

* No history of CRS
* SNOT-20 score <1.0
* No evidence of sinus disease on preoperative imaging

Exclusion Criteria:

* Control patients with any evidence of CRS, by history, survey, or imaging criteria would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04-30 (Actual); Study Completion 2008-04-30 (Actual)

PRIMARY OUTCOMES:
Microbial community profiling using the PhyloChip, MycoChip, and ViroChip will yield vast quantities of data to be reduced in dimensions for interpretation. Pathogens detected in the nasal mucus of patients with CRS will be compared to healthy controls. | Immediate Preoperative period.

SECONDARY OUTCOMES:
The presence or absence of a given microorganism will be compared to previously published data obtained using either traditional culture methods or other genomic methods. | Immediate preoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Goldberg, MD, MSCE, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Dept of Otolaryngology-HNS, San Francisco, California, United States